CLINICAL TRIAL: NCT00573937
Title: Methadone Versus Morphine for Moderate to Severe Cancer-Related Pain: A Double-Blind Randomized Parallel Group Study
Brief Title: Methadone Versus Morphine for Cancer-Related Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Donald W. Northfelt, M.D., MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-003051
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2010-11-04 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Neoplasms; Pain
Keywords: Neoplasms; Pain; Methadone; Morphine
MeSH Terms: conditions — Neoplasms; Pain | interventions — Methadone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone (Active Comparator): Oral methadone 2.5 mg every 8 hours, and oral methadone 2.5 mg every 4 hours as needed for breakthrough pain.
  Interventions: Drug: Methadone
- Morphine (Active Comparator): Oral slow-release morphine (15 mg) every 8 hours, and immediate-release morphine (10 mg) every 4 hours as needed for breakthrough pain.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — Oral methadone 2.5 mg every 8 hours, and oral methadone 2.5 mg every 4 hours as needed for breakthrough pain.
  Other Names: Methadone Hydrochloride; Methadose; Dolophine Hydrochloride
  Arms: Methadone
Drug: Morphine — Oral slow-release morphine 15 mg every 8 hours, and oral immediate-release morphine 10 mg every 4 hours as needed for breakthrough pain.
  Other Names: Morphine Sulfate
  Arms: Morphine

SUMMARY:
The purpose of this study is to compare methadone with morphine in the management of moderate to severe cancer pain.

DETAILED DESCRIPTION:
Treatment of cancer pain is based on the World Health Organization (WHO) step ladder approach to the use of analgesic drugs. Medication potency increases at each step of the WHO ladder, from nonopioid (step 1; e.g., aspirin and nonsteroidal anti-inflammatory drugs) through weak opioids (step 2; e.g. codeine) plus a nonopioid to strong opioids (step 3; e.g., morphine) plus a nonopioid analgesic. Morphine is considered the gold standard for the treatment of moderate to severe pain, but this is based on level C criteria. Research has discovered that methadone is a potent opioid that operates at several levels which are important for pain control. The primary aim is to compare morphine versus methadone as a first-line analgesic in patients with moderate to severe cancer pain. Patients will be randomized to receive either oral slow-release morphine (15 mg) every 8 hours and immediate-release morphine (10 mg) every 4 hours as needed for breakthrough pain or oral methadone 2.5 mg every 8 hours and methadone 2.5 mg every 4 hours as needed for breakthrough pain. Our hypothesis is that methadone will provide equivalent pain control efficacy after 4 weeks of therapy. We postulate that methadone will be as preferable as morphine as an analgesic. We will compare the two drugs via adverse effects and compare stability of analgesia via comparison of the number of breakthrough pain episodes. The study will attempt to establish equivalency of methadone as a first-line analgesic for moderate to severe cancer pain.

ELIGIBILITY:
Inclusion Criteria:

* Must have a telephone
* Age: patient must be 18 years or older and less than 70 years of age
* Life expectancy of 3 months or greater
* No prior use of step-3 opioids (step 2 opioids are allowed)
* Provision of informed consent
* Score of 26 or greater on Mini-Mental Status Exam (MMSE) (to be done by investigator if there is question about mental status)
* Nonmalignant pain will be excluded; however, if the patient has both malignant and nonmalignant pain, entry into the trial will be determined by the predominant site of pain
* Moderate to severe cancer related pain that requires the use of step-3 opioids
* Normal renal function
* There will be no exclusionary criteria based on Karnofsky score
* Must live no more than 1 hour away from clinic
* Patient must have pain severity of 5-7/10 on a 0-10 pain scale

Exclusion Criteria:

* Nursing home patients
* Obvious cognitive dysfunction
* Intractable nausea or vomiting
* A true allergy or intolerance to opioids
* Unstable renal function
* Undergoing therapeutic procedures likely to influence pain during the study period
* Gastrointestinal pathology or surgery that influences absorption of morphine or methadone
* Must not have had treatment with radiotherapy, chemotherapy or radionuclides in the last 30 days
* History of drug seeking behavior
* Respiratory compromise
* Treatment with bisphosphonates within the last month
* Use of MAO inhibitors
* Drugs that interfere with CYP34A or CYP2D6
* Drugs that interfere with morphine metabolism
* Retroviral therapies
* Active radiation or antineoplastic therapies
* Hepatic dysfunction
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study
* Study will exclude women who are pregnant and/or nursing
* Women who are of child bearing potential must have a negative urine pregnancy test
* Patients with a recent substance abuse history will be excluded
* Patients with major depression will be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Northfelt, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the outpatient hematology/oncology clinic, inpatient cancer service, and palliative care unit, at a tertiary medical center from September 2007 to April 2009.
Pre-assignment Details: One subjects was assigned to standard control treatment. No subjects received the experimental treatment. No subject data were analyzed.
Period: Overall Study
Arm/Group | Methadone | Morphine
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Study Terminated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone | Morphine | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 48 | 48
Gender [Number; unit: participants]
  Female |  | 1 | 1
  Male |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Numeric Pain Scale Score
Description: Subjects will be verbally questioned about their pain on a scale from 0 to 10, with 0 being symptoms are absent to 10, the worst possible pain. Response to treatment is defined as a 33% reduction in pain score from the baseline to the Week 4 pain score.
Time Frame: Baseline, Week 4
Population: Due to slow accrual, the study was terminated and no data were analyzed.
Arm/Group | Methadone | Morphine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Numeric Pain Scale Score
Description: Subjects will be verbally questioned about their pain on a scale from 0 to 10, with 0 being symptoms are absent to 10, the worst possible pain.
Time Frame: 48 hours
Population: Due to slow accrual, the study was terminated and no data were analyzed.
Arm/Group | Methadone | Morphine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 4 weeks
Arm/Group | Methadone | Morphine
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Due to slow accrual of subjects, the study was terminated after one subject started in the standard control group (morphine). No subject received investigational study drug (methadone). Therefore no data were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes